CLINICAL TRIAL: NCT00316498
Title: A Phase I/II Randomized, Controlled Study of OGT 918 in Adult and Juvenile Patients With Niemann Pick C Disease
Brief Title: Saccadic Eye Movements in Patients With Niemann-Pick Type C Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030011; 03-EI-0011
Record Dates: First submitted 2006-04-19; First posted 2006-04-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Niemann Pick Diseases
Keywords: Eye Movement; Niemann Pick C
MeSH Terms: conditions — Niemann-Pick Diseases | interventions — miglustat

INTERVENTIONS:
Drug: OGT918

SUMMARY:
This study is done in conjunction with a trial, conducted at Columbia University College of Physicians and Surgeons in New York and the Royal Manchester Children's Hospital in England, to examine the effectiveness of a new drug called OGT 918 for treating Niemann-Pick Type C (NPC) disease. Patients with this genetic disorder do not transport lipids (fatty substances) in their cells, resulting in problems of the liver, spleen and brain. An early sign of NPC is a reduced ability to move the eyes rapidly up and down or from side to side. These voluntary eye movements are called saccades. Patients in the OGT 918 trial who participate in this sub-study will have their saccadic eye movements measured to see if improvement occurs with OGT 918 treatment.

Patients with Niemann-Pick Type C disease 12 years of age and older who are enrolled in the OGT 918 trial described above may be eligible for this study.

Participants will have both vertical (up and down) and horizontal (side to side) saccadic eye movements measured at two time points before starting treatment with OGT 918 and after 12 months of treatment. For the test, patients sit in a chair with their head positioned as for a regular eye examination (steadied by a chin cup and headrest) and follow with their eyes a series of lights or laser spots moving on a screen at a distance of 1 meter (3 feet). During the test, patients wear either special recording glasses, infrared goggles, or special contact lenses for measuring eye movements. A full eye evaluation lasts about 1 hour, and each eye is evaluated twice. The evaluations are separated in time by at least an hour, and possibly a day.

DETAILED DESCRIPTION:
None given, verified by PI.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with NPC disease confirmed by abnormal cholesterol esterification and abnormal filipin staining.

Patients aged 12 and over. Body weight must not be less than 14 kg.

Patients who can ingest a capsule.

EXCLUSION CRITERIA:

Patients younger than 18 who are unable to give informed assent and/or whose legal guardian is unable to provide informed consent.

Patients aged 18 and over who cannot provide informed consent and/or whose legal guardian is unable to provide witnessed informed consent.

Fertile patients who do not agree to use adequate contraception throughout the study and for three months after cessation of OGT 918 treatment.

Patients who cannot tolerate the study procedures or who are unable to travel to the study center as required by this protocol.

Patients currently undergoing therapy with other investigational agents or patients taking drugs or food supplements which may interfere with gastrointestinal absorption or motility.

Patients suffering from clinically significant diarrhoea (greater than 3 liquid stools per day for greater than 7 days) without definable cause within 3 months of Screening Visit, or who have a history of significant gastrointestinal disorders.

Patients with an intercurrent medical condition that would render them unsuitable for the study e.g. HIV, hepatitis infection.

Patients who in the opinion of the investigator (for whatever reason) are thought to be unsuitable for the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2002-10-17; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Columbia University, New York, New York
- Oxford GlycoSciences Ltd., Abingdon, United Kingdom

REFERENCES:
- [Background] Platt FM, Neises GR, Reinkensmeier G, Townsend MJ, Perry VH, Proia RL, Winchester B, Dwek RA, Butters TD. Prevention of lysosomal storage in Tay-Sachs mice treated with N-butyldeoxynojirimycin. Science. 1997 Apr 18;276(5311):428-31. doi: 10.1126/science.276.5311.428. PMID 9103204